CLINICAL TRIAL: NCT06326515
Title: Cognitive Behavior Therapy for Depression, Stigmatization, Criminogenic Cognition, and Quality of Life Among Patients With Opioid Use Disorder (OUD): A Randomized Control Trial
Acronym: CBT with OUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Qasir Abbas, Principle Investigator, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Government College University
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Psychoeducation
Keywords: Opioid use disorder, Cognitive behaviour therapy, Primary symptoms, Secondary symptoms
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cognitive Restructuring

STUDY DESIGN:
Intervention Model Description: Randomized control trial design would be used in this study. It would be two arm study and there would be two groups an experimental and wait-list control group. Experimental group will receive intervention and another group would be placed in waitlist. In this research, parallel group design would be used. We will give treatment to all participants in a parallel way. Allocation ratio and framework would be equivalence i.e., treatment group and control group would be equal number of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Treatment Group (Experimental): Experimental: Treatment Group
  Experimental Group:
  Participants in the experimental group would receive 8-10 session of psychoeducational based Program.
  Waitlist control Group:
  Participants in the Control group would not receive psychoeducational Intervention
  Interventions: Behavioral: psychoeducation; Behavioral: Stigma Reduction and Relapse Management
- No Intervention: Control Group (No Intervention): No Intervention: Control Group
  Control Group:
  Participants in the control group did not receive the said psychoeducational intervention

INTERVENTIONS:
Behavioral: psychoeducation — To identify and recognize the cognitive distortions To explore the automatic thoughts and emotions about illness Evaluate and respond to thoughts, emotions, and beliefs Automatic thought records were used by patients with some help from therapist (Chattopadhyay et al., 2017).
  The cognitive errors were corrected using individual cognitive strategies (Chattopadhyay et al., 2017).
  Other Names: Cognitive Conceptualization and Cognitive Restructuring
  Arms: Experimental: Treatment Group
Behavioral: Stigma Reduction and Relapse Management — To improve ability to effectively cope with lapse and relapse (Brown & Vanable, 2008).
  To improve relapse management skills (Brown & Vanable, 2008). Emphasized skill development to cope with OUD-related stressors (Zhang, 2021). To change their conception of OUD (Tshabalala & Visser, 2011). To change their sense of self-worth and to empower them with more adaptive ways of thinking (Tshabalala & Visser, 2011).
  To deal with their experience of stigma (Tshabalala & Visser, 2011).
  Arms: Experimental: Treatment Group

SUMMARY:
to investigate the impact of cognitive behavior therapy for psychiatric problems among patients with opioid use disorder with relapse condition.

In this randomize control trail (RCT), N=120 patients with relapse condition would be taken. After enrolment patients' eligibility assessment would be completed and then n=60 patients would be allocated to experimental (n=30) and waitlist control (n=30) through random assignment. Patient's age range would be between 20 to 30 years.

DETAILED DESCRIPTION:
Background: Opioid use disorder causes severe mental health problems with high mortality and morbidity (Harford, Yi, & Grant, 2013). Cognitive behavior therapy is found an evidence-based treatment modality to address psychiatric problems among individuals with substance use disorders (Cosci et al., 2007).

Objectives: to investigate the impact of cognitive behavior therapy for psychiatric problems among patients with opioid use disorder with relapse condition.

Hypothesis: After review of literature, cognitive behavior therapy would reduce criminogenic cognition, depressive symptoms, stigma and addiction severity and will improve coping strategies and the quality of life between experimental and waitlist control.

Methods: In this randomize control trail (RCT), N=120 patients with relapse condition would be taken. After enrolment patients' eligibility assessment would be completed and then n=60 patients would be allocated to experimental (n=30) and waitlist control (n=30) through random assignment. Patient's age range would be between 20 to 30 years.

Measures: Demographic form and in-depth clinical interview would be used conducted to take history of the participants' problems. Moreover, Alcohol, Smoking and Substance Involvement Screening Test (ASSIST; Henry-Edwards et al., 2003; Hussain et al., 2022), Criminogenic Cognition Scale (CCS;Tangney, at el, 2012; Jamil & Fatima, 2018) Perceived Stigma of Addiction Scale (PSAS; Luoma et al, 2010; Shahzad et al., 2021), Patient Health Questionnaire (PHQ-9; Robert et al. 1999; Ahmad et al, 2018), Relapse Risk Scale (RRS; Marlatt & Gordon, 1985; Hussain et al., 2016), Brief Cope Inventory (BCI; Carver, 1997; Shahzad et al., 2020) and World Health Organization Quality-of-Life Scale (WHOQOL; WHO, 2004; Khalid & Kausar, 2006) would be used as secondary measures.

Interventions: The treatment protocol would be prepared on the base of CBT with specific goals including short term and long term. 8-12 therapeutic sessions would be given with twice a week interval in one-on-one sitting.

Procedure: After approval from the BOS and Advance Studies and Research (ASR), G. C. University Faisalabad, study proposal would be submitted in the Institutional Review Board (IRB), G. C. University Faisalabad for further approval. Furthermore, study protocol would be registered in WHO recognised registry for further approval to conduct RCT. Then data would be collected after getting consent from the institutions as well as from the participants. In RCT, participants eligibility assessment would be completed after enrolment then they will be allocated to experimental and control groups through random assignment. CBT based 8-12 therapeutic sessions would be given with twice a week interval in one-on-one sitting.

Statistical analysis: Study-I: Descriptive statistics (i.e., M, SD & f) will be used to calculate demographic characteristics of the sample. Correlation statistics, t-test, and mediation analysis using PROCESS would be used. Study-II: Descriptive statistics (i.e., M & SD), chi-square statistics, power analysis, and repeated measure ANOVA statistics would be used. All statistical computation would be calculated by using SPSS 26.0. sample size would be calculated using G-Power Software.

ELIGIBILITY:
Inclusion Criteria:

In this study, only patients they have history of relapse would be taken. Patient's age range would be between 20 to 30 years. Patients would be taken who are un-married and belong from middle social economic status. Participants would be diagnosed according to the DSM-V.

-

Exclusion Criteria:

Participants with more than 4-time history of relapse and more than 5 years of history of illness would be excluded from the study. Participants with different medical comorbidities, and intellectual disability would be excluded. Participants who would not sign the consent form or would not complete all the research procedures would also exclude from the study.

-

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST; Henry-Edwards et al., 2003; Hussain et al., 2022). | 1-2 weeks
  It was developed by the World Health Organization (WHO) and adopted by Hussain et al. (2022) to screen out people's use of psychoactive substances.
Criminogenic Cognition Scale (CCS;Tangney, at el, 2012; Jamil & Fatima, 2018): | after Allocation 1 week
  measure that has been reported to have statistically sound psychometric properties (Tangney etal., 2012). The 25 item Criminogenic Cognitions Scale (CCS) was designed to tap 5 dimensions
Patient Health Questionnaire (PHQ-9; Robert et al. 1999; Ahmad et al, 2018). | after Allocation 1 week
  It is a depression screening instruments that can be self-administered.
Relapse Risk Scale (RRS; Marlatt & Gordon, 1985; Hussain et al., 2016): | after Allocation 1 week
  The RRS was developed by Marlatt and Gordon (1985) and adopted by Hussain et al. (2016) to assess the cognitive and behavioral triggers toward relapse.
Perceived Stigma of Addiction Scale | after Allocation 1 week
  The PSAS developed by Luoma et al. (2010) and adopted by Shahzad et al. (2021) to assess perceived stigma among substance users and patients with OUD specifically.
Brief Cope Inventory (BCI) | after Allocation 1 week
  The Brief COPE is a 28-item multidimensional measure of strategies used for coping or regulating cognitions in response to stressors

SECONDARY OUTCOMES:
World Health Organization Quality-of-Life Scale | after Allocation 1 week
  it assesses impact of negative events on subjective well-being across four areas of an individual's life that is, physical, psychological, social, and environmental domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Khalid Mahmood, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No